CLINICAL TRIAL: NCT02953015
Title: Effects of Cervical and Thoracic Manipulative Techniques Combined With OnabotulinumtoxinA Prophylaxis in the Management of Chronic Migraine: a Pilot Single-blind Randomized Controlled Trial
Brief Title: Non-pharmacological Management of Chronic Migraine
Acronym: MIGRANE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universita di Verona (Other)
Collaborators: Marialuisa Gandolfi (Unknown)
Responsible Party: Principal Investigator, Nicola Smania, MD, Clinical Professor, MD, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIGRANE
Record Dates: First submitted 2016-09-19; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Headache
Keywords: Chronic Migraine; Manipulative treatments; Transcutaneous Electrical Nerve Stimulation
MeSH Terms: conditions — Headache | interventions — Transcutaneous Electric Nerve Stimulation; Electric Stimulation; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manipulative articulatory and myofascial techniques Group (Experimental): Manipulative and myofascial techniques
  Interventions: Behavioral: Manipulative articulatory (ART) and myofascial techniques; Drug: OnabotulinumtoxinA (Prophylaxis therapy)
- Transcutaneous Electrical Nerve Stimulation Group (Active Comparator): Electrical Nerve Stimulation
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation; Drug: OnabotulinumtoxinA (Prophylaxis therapy)

INTERVENTIONS:
Behavioral: Manipulative articulatory (ART) and myofascial techniques — Three manipulative articulatory (ART) and myofascial techniques will be performed to improve cervical and thoracic spine joint mobility and reducing soft tissue stiffness in the cervico-thoracic spine. ART technique is a low velocity to high amplitude technique where each joint is carried through its full motion to increase range of movement. The activating force is either a repetitive springing motion or repetitive concentric movement of the joint through the restrictive barrier. Myofascial technique is directed at the muscle and fascia treatment. It engages continual palpatory feedback to achieve release of myofascial tissues. During each treatment session, each technique will be carried out for 10 minutes including 2 minutes of resting.
  Other Names: Manipulations
  Arms: Manipulative articulatory and myofascial techniques Group
Device: Transcutaneous Electrical Nerve Stimulation — Transcutaneous Electrical Nerve Stimulation (TENS) of the upper trapezius muscle will be applied by a portable machine Master 932 (Elettronica Pagani SRL, Milan, Italy) that generates symmetric, bi-phasic rectangular pulses with 140μ sec duration. The current frequency will be set at 150 Hz and intensity will be increased up to patient's perception of paresthesia. The negative electrode will be placed on the active TrPs of the upper trapezius muscle and the positive one was on acromial tendon insertional site. The total duration of each application will be 20 minutes. Treatment frequency and duration will be the same of the EG treatment (1 session/week for 4 weeks). Each session will consist of 20 min of TENS and 10 min of resting in sitting position with the head lean on a pillow.
  Other Names: Electrical stimulations
  Arms: Transcutaneous Electrical Nerve Stimulation Group
Drug: OnabotulinumtoxinA (Prophylaxis therapy) — Prophylaxis therapy with OnabotulinumtoxinA according to the PREEMPT protocol (155U every three months into 31 injection site).
  Other Names: OnabotulinumtoxinA injections

SUMMARY:
Chronic migraine (CM) is a very disabling disorder with grave socioeconomic consequences. Pharmacological approaches can affect mechanisms of pain production, while rehabilitation such as Transcutaneous Electrical Nerve Stimulation and Manual Therapy may reduce the neuromuscular contributing factors. The main aim of the study is to evaluate the effects of cervical and thoracic manipulative techniques combined with OnabotulinumtoxinA prophylaxis on headache frequency in patients with Chronic Migraine (CM). The second aim is to evaluate the training effects on the intensity of headache attacks, analgesic consumption, cervical range of motion, TrPs sensitivity and disability. The hypothesis is that the manipulative treatment would alleviate CM symptoms and, in turn, decrease the analgesic consumption.

DETAILED DESCRIPTION:
The present study is a single-blind randomized controlled trial conducted according to the Declaration of Helsinki, the guidelines for Good Clinical Practice, and the Consolidated Standards of reporting Trials (CONSORT) Statement guidelines. The examiner will be blinded to group assignment. If eligible, patients will be allocated to the experimental group (EG) or the control group (CG) using an automated randomization system (Allocation ratio 1:1). The group allocation will be kept concealed by means of sealed numbered envelopes. The randomization list was locked in a desk drawer accessible only to the main investigator. All the treatments and assessment will be performed in the Neurorehabilitation Unit of Azienda Ospedaliera Universitaria Integrata of Verona (Italy).

Patients will be asked to complete a daily headache diary, which is routinely administered to all patients with CM admitted at our Unit for OnabotulinumtoxinA prophylaxis. In the context of this study, daily headache diaries during 1 month pre-treatment (T0), during the treatment (treatment phase) and 1 month post-treatment (T1) will be considered.

Moreover, at T0 a questionnaire concerning clinical and demographic data as well as some habits like consumption of coffee and alcohol, and smoking will be administered. According to the nature of the study feasibility and efficacy outcomes will be defined. Feasibility outcomes were the patients' compliance during treatments, any adverse events (i.e. pain, discomfort) occurred during the treatment, and the number of training session performed. Primary and secondary outcome measures will be categorized as efficacy outcomes.

ELIGIBILITY:
Inclusion criteria will be:

* age between 18 and 65 years;
* diagnosis of CM according to fhe International Classification of Headache Criteria-III;
* ineffective assumption of at least 3 different drug classes recommended by the international guidelines of migraine treatment;
* intolerance to/inefficacy of primary prophylaxis therapy;
* prophylactic treatment with OnabotulinumtoxinA according to the Phase III Research Evaluating Migraine Prophylaxis Therapy (PREEMPT) protocol;
* at least two consecutive OnabotulinumtoxinA injections.

Exclusion criteria will be:

* contraindications to onaBoNTA injection;
* presence of other neurologic disorders that can cause/sustain migraine;
* onaBoNTA treatment for purposes other than those of this study;
* other non-pharmacological treatments for migraine (e.g. massage, acupuncture);
* severe and unstable cardiovascular and cerebrovascular disease;
* presence of infections, psychiatric diseases or functional disorders in any head structure;
* severe osteoporosis;
* vertebral or arm fractures; alcohol/drug abuse;
* relevant medical therapy changes during the trial;
* incomplete headache diaries with missing information.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the number of days without headache | Baseline, 1 month
  Time frame: from date of randomization up to 1 months.

SECONDARY OUTCOMES:
Total time with headache (hrs) | Baseline, 1 month
  Time frame: from date of randomization up to 1 months.
Headache intensity reported as mild, moderate and severe per month. | Baseline, 1 month
  Time frame: from date of randomization up to 1 months.
Average duration of attacks (hrs) | Baseline, 1 month
  Time frame: from date of randomization up to 1 months.
The analgesic consumption reported as the number of total acute analgesic (NSAIDs/Triptans), NSAID and Triptans per month. | Baseline, 1 month
  Time frame: from date of randomization up to 1 months.
Cervical Active Range of Motion (Degrees) | Baseline, 1 month
  Time frame: from date of randomization up to 1 months.
Headache Impact Test-6 (HIT-6). | Baseline, 1 month
  Time frame: from date of randomization up to 1 months.
Migraine Disability Assessment Scale (MIDAS). | Baseline, 1 month
  Time frame: from date of randomization up to 1 months.
Trigger points sensitivity (lbf/kgf or kgf/N) | Baseline, 1 month
  Trigger point sensitivity will be assessed by measuring the pressure pain threshold (PPT) with a Wagner algometer 162 (Wagner Instruments, Riverside, CT, USA). The PPT corresponds to the force needed to induce a difference between a feeling of simple pressure and a painful sensation. PPT assessment will be performed on the frontalis, temporalis and occipitalis, and upper trapezius muscles.
  Time frame: from date of randomization up to 1 months.
Number of patients that withdrawn the study (dropouts), and patients reporting side effects | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Smania, MD, Principal Investigator — Universita di Verona
Locations (1):
- University of Verona, Verona, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buse DC, Manack AN, Fanning KM, Serrano D, Reed ML, Turkel CC, Lipton RB. Chronic migraine prevalence, disability, and sociodemographic factors: results from the American Migraine Prevalence and Prevention Study. Headache. 2012 Nov-Dec;52(10):1456-70. doi: 10.1111/j.1526-4610.2012.02223.x. Epub 2012 Jul 25. PMID 22830411